CLINICAL TRIAL: NCT01617226
Title: Phase II Randomised Trial of 5-azacitidine Versus 5-azacitidine in Combination With Vorinostat in Patients With Acute Myeloid Leukaemia or High Risk Myelodysplastic Syndromes Ineligible for Intensive Chemotherapy
Brief Title: Randomised Study of Azacitidine Versus Azacitidine With Vorinostat in Patients With AML or High Risk MDS
Acronym: RAvVA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Leukemia Research Fund (Other); Celgene (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Professor Charles Craddock, Professor of Haemato-Oncology, Director of Stem Cell Transplant Unit and Transitional Director of Birmingham Health Partners, University of Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG_11-187
Record Dates: First submitted 2012-06-06; First posted 2012-06-12 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- azacitidine (Active Comparator): azacitidine (75mg/m2) by SC injection on 7 consecutive days (excluding weekends), starting day 1 of 28-day cycles for up to 6 cycles. This should be delivered in a 5-2-2 schedule
  Interventions: Drug: Azacitidine
- azacitidine and vorinostat (Active Comparator): Patients will receive (75mg/m2) azacitidine by SC injection on 7 consecutive days (excluding weekends), starting day 1 of 28-day cycles for up to 6 cycles. Azacitidine should be delivered in a 5-2-2 schedule. Vorinostat (300mg bid) will be taken orally for 7 consecutive days starting on day 3 of each cycle in 28-day cycles for up to 6 cycles. (Day 3 is defined as the 3rd day of azacitidine administration).
  Interventions: Drug: Azacitidine; Drug: Vorinostat

INTERVENTIONS:
Drug: Azacitidine — Azacitidine both arms; 75mg/m^2 by subcutaneous injection for 7 days of a 28-day cycle for up to 6 cycles.
  Other Names: vidaza, ATC code L01BC07, cas number 320-67-2
Drug: Vorinostat — Vorinostat (with azacitidine) combined therapy arm; 300mg twice daily for 7 days starting on day 3 of each cycle in 28-day cycles for up to 6 cycles.
  Other Names: MK-0683, ATC code L01XX38, cas number 149647-78-9
  Arms: azacitidine and vorinostat

SUMMARY:
This is a multicentre, open-label, randomised phase II trial comparing azacitidine monotherapy with combined azacitidine and vorinostat in patients with newly diagnosed, relapsed or refractory acute myeloid leukaemia or high risk myelodysplastic syndromes ineligible for intensive chemotherapy.

DETAILED DESCRIPTION:
Acute Myeloid Leukaemia (AML) is a common haematological malignancy. As a result of improvements in myelosuppressive chemotherapy and stem cell transplantation, the outcome of children and young adults with AML has improved substantially in the past three decades. By contrast there has only been limited progress in the development of new treatments for older adults in whom long term survival is less than 20% at present.

There is an urgent need to develop more effective treatment options for the treatment of AML and high risk MDS in older adults. Accumulating evidence suggests that Azacitidine is a potentially important treatment modality in newly diagnosed, relapsed/refractory AML and high risk MDS. Phase II trials in AML and MDS demonstrate increased clinical activity of azacitidine when combined with a HDACi. However no randomised trials have yet examined the important question of whether concurrent HDACi administration increases the clinical activity of Azacitidine. Vorinostat is a new HDACi which shows significant clinical activity in combination with Azacitidine in patients with AML and MDS.

We therefore propose a randomised trial of azacitidine compared with azacitidine and vorinostat combination therapy in older adults with newly diagnosed, relapsed, refractory AML or high risk MDS ineligible for intensive chemotherapy. This will represent the first randomised trial, addressing whether there is a clinical benefit to be gained from combining treatment with azacitidine with a HDACi in patients with newly diagnosed, relapsed, refractory AML or high risk MDS for whom limited therapeutic options currently exist.

ELIGIBILITY:
Inclusion Criteria:

- Adults with AML (except Acute Promyelocytic Leukaemia (APL)) as defined by the World Health Organisation (WHO) Classification or patients with high risk MDS categorised as INT-2 or high risk according to the International Prognostic Scoring System (IPSS) who are deemed ineligible for intensive chemotherapy on the grounds of age or co-morbidities with ONE of the following disease status:- i) Newly diagnosed OR

ii) Relapsed Disease: patients must have achieved a previous morphological CR and show evidence of recurrent disease OR

iii) Refractory Disease: patients who have failed to achieve a morphological CR with previous therapy

* Patients are able to receive treatment as out-patient
* Adequate renal and hepatic function as defined in the Protocol
* Patients have given written informed consent
* ECOG performance status less than or equal to 2

Exclusion Criteria:

* Patients with greater than class III NYHA cardiac impairment
* Blastic transformation of Chronic Myeloid Leukaemia
* Prior allogeneic/autologous haematopoietic stem cell transplant
* Pregnant or lactating women
* Adults of reproductive potential not willing to use appropriate, effective, contraception during the trial and for specified amount of time afterwards
* Patients who have received prior histone deacetylase inhibitor (HDACi) treatment as anti-tumour therapy. (Patients who have received HDACi treatment for other indications e.g valproic acid for epilepsy may enrol after a 30-day washout period)
* Previous anti-tumour therapies, including prior experimental agents or approved anti-tumour small molecules and biologics, within 30 days before the start of protocol treatment. (Patients receiving anti-tumour therapies to control blood counts may enrol into the trial)
* Patients who have received prior treatment with demethylating agents such as 5-azacitidine or decitabine
* Patients with contraindications to receiving azacitidine or vorinostat such as hypersensitivity, patients unable to have a subcutaneous injection or swallow oral capsules
* Active symptomatic fungal, bacterial, and/or viral infection including known active HIV or known viral (A, B, or C) hepatitis
* Any co-morbidity that could limit compliance with the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2012-09; Primary Completion 2016-03 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Phase II - Overall Response Rate | Upto 6 months
  Patients are expected to receive 6 cycles of treatment which is expected to be completed over a period of 6 months. Each cycle lasts for 28 days. Overall response rate (CR, CRi, PR) as defined by Cheson criteria will be assessed during this time. This will be measured for all patients receiving treatment recruited over a 24 month period.
Phase II - Overall Survival | Up to 24 months
  Overall survival is defined as the time from date of randomisation to the date of death from any cause. Patients discontinuing study, lost to follow up or still alive at the end of the study (up to 24 months) will be censored at the date of last follow-up.

SECONDARY OUTCOMES:
Phase II - Toxicities measured by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) | Up to 28 days
  Toxicities will be measured and graded according to the NCI CTCAE v4 from the date of randomisation until 28 days following treatment discontinuation over the duration of the follow up period which is 24 months.
Phase II - Complete Remission (CR) within 6 cycles of treatment | Up to 6 months
  Complete remission within 6 cycles of treatment as defined by Cheson criteria will be assessed. It is expected patients will receive 6 cycles of treatment, which is expected to be completed over a period of 6 months, as each cycle is 28 days. This will be measured for all patients receiving treatment recruited over a 24 month period.
Phase II - Duration of response | Up to 24 months
  This will be measured from date of documented response until date of documented progression, assessed for up to 24 months.
Phase II - Dose intensity | Up to 24 months
  Dose intensity defined as the total dose prescribed to each patient as a proportion of the protocol dose. This will measured for each patient receiving treatment, assessed up to 24 months.
Phase II - Quality of Life measured by questionnaires | Up to 24 months
  Quality of Life will be measured using the EORTC QLQ-C30 and EuroQol EQ-5D-5L questionnaires. This will be measured for each patient receiving treatment until end of treatment, assessed for up to 24 months.
Phase II - Medical Resource Use | Up to 24 months
  Medical resource use is defined in terms of days in hospital, blood product usage and days on anti-biotics and will be measured from date of randomisation until 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Charles F Craddock, Professor, Principal Investigator — University of Birmingham
Locations (13):
- United Kingdom (13):
  - Barts and the London NHS Trust, London, Greater London
  - King's College Hospital, London, Greater London
  - Hammersmith Hospital, London, Greater London
  - The Christie Hospital, Manchester, Greater Manchester
  - Royal Liverpool University Hospital, Liverpool, Merseyside
  - Belfast City Hospital, Belfast, Northern Ireland
  - Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire
  - Oxford University Hospitals NHS Trust, Oxford, Oxfordshire
  - University Hospital of Wales, Cardiff, South Wales
  - Queen Elizabeth Hospital, Birmingham, West Midlands
  - St James's University Hospital, Leeds, West Yorkshire
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Southampton General Hospital, Southampton

REFERENCES:
- [Background] Cheson BD, Bennett JM, Kopecky KJ, Buchner T, Willman CL, Estey EH, Schiffer CA, Doehner H, Tallman MS, Lister TA, Lo-Coco F, Willemze R, Biondi A, Hiddemann W, Larson RA, Lowenberg B, Sanz MA, Head DR, Ohno R, Bloomfield CD; International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia. Revised recommendations of the International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia. J Clin Oncol. 2003 Dec 15;21(24):4642-9. doi: 10.1200/JCO.2003.04.036. PMID 14673054
- [Background] Dohner H, Estey EH, Amadori S, Appelbaum FR, Buchner T, Burnett AK, Dombret H, Fenaux P, Grimwade D, Larson RA, Lo-Coco F, Naoe T, Niederwieser D, Ossenkoppele GJ, Sanz MA, Sierra J, Tallman MS, Lowenberg B, Bloomfield CD; European LeukemiaNet. Diagnosis and management of acute myeloid leukemia in adults: recommendations from an international expert panel, on behalf of the European LeukemiaNet. Blood. 2010 Jan 21;115(3):453-74. doi: 10.1182/blood-2009-07-235358. Epub 2009 Oct 30. PMID 19880497
- [Background] Fenaux P, Mufti GJ, Hellstrom-Lindberg E, Santini V, Gattermann N, Germing U, Sanz G, List AF, Gore S, Seymour JF, Dombret H, Backstrom J, Zimmerman L, McKenzie D, Beach CL, Silverman LR. Azacitidine prolongs overall survival compared with conventional care regimens in elderly patients with low bone marrow blast count acute myeloid leukemia. J Clin Oncol. 2010 Feb 1;28(4):562-9. doi: 10.1200/JCO.2009.23.8329. Epub 2009 Dec 21. PMID 20026804
- [Background] Sudan N, Rossetti JM, Shadduck RK, Latsko J, Lech JA, Kaplan RB, Kennedy M, Gryn JF, Faroun Y, Lister J. Treatment of acute myelogenous leukemia with outpatient azacitidine. Cancer. 2006 Oct 15;107(8):1839-43. doi: 10.1002/cncr.22204. PMID 16967444
- [Background] Soriano AO, Yang H, Faderl S, Estrov Z, Giles F, Ravandi F, Cortes J, Wierda WG, Ouzounian S, Quezada A, Pierce S, Estey EH, Issa JP, Kantarjian HM, Garcia-Manero G. Safety and clinical activity of the combination of 5-azacytidine, valproic acid, and all-trans retinoic acid in acute myeloid leukemia and myelodysplastic syndrome. Blood. 2007 Oct 1;110(7):2302-8. doi: 10.1182/blood-2007-03-078576. Epub 2007 Jun 27. PMID 17596541
- [Background] Jabbour E, Giralt S, Kantarjian H, Garcia-Manero G, Jagasia M, Kebriaei P, de Padua L, Shpall EJ, Champlin R, de Lima M. Low-dose azacitidine after allogeneic stem cell transplantation for acute leukemia. Cancer. 2009 May 1;115(9):1899-905. doi: 10.1002/cncr.24198. PMID 19235255
- [Background] de Lima M, Giralt S, Thall PF, de Padua Silva L, Jones RB, Komanduri K, Braun TM, Nguyen HQ, Champlin R, Garcia-Manero G. Maintenance therapy with low-dose azacitidine after allogeneic hematopoietic stem cell transplantation for recurrent acute myelogenous leukemia or myelodysplastic syndrome: a dose and schedule finding study. Cancer. 2010 Dec 1;116(23):5420-31. doi: 10.1002/cncr.25500. Epub 2010 Jul 29. PMID 20672358
- [Background] Garcia-Manero G, Yang H, Bueso-Ramos C, Ferrajoli A, Cortes J, Wierda WG, Faderl S, Koller C, Morris G, Rosner G, Loboda A, Fantin VR, Randolph SS, Hardwick JS, Reilly JF, Chen C, Ricker JL, Secrist JP, Richon VM, Frankel SR, Kantarjian HM. Phase 1 study of the histone deacetylase inhibitor vorinostat (suberoylanilide hydroxamic acid [SAHA]) in patients with advanced leukemias and myelodysplastic syndromes. Blood. 2008 Feb 1;111(3):1060-6. doi: 10.1182/blood-2007-06-098061. Epub 2007 Oct 25. PMID 17962510
- [Background] Khanim FL, Bradbury CA, Arrazi J, Hayden RE, Rye A, Basu S, MacWhannell A, Sawers A, Griffiths M, Cook M, Freeman S, Nightingale KP, Grimwade D, Falciani F, Turner BM, Bunce CM, Craddock C. Elevated FOSB-expression; a potential marker of valproate sensitivity in AML. Br J Haematol. 2009 Feb;144(3):332-41. doi: 10.1111/j.1365-2141.2008.07449.x. Epub 2008 Nov 22. PMID 19036090
- [Background] Wijermans P, Lubbert M, Verhoef G, Bosly A, Ravoet C, Andre M, Ferrant A. Low-dose 5-aza-2'-deoxycytidine, a DNA hypomethylating agent, for the treatment of high-risk myelodysplastic syndrome: a multicenter phase II study in elderly patients. J Clin Oncol. 2000 Mar;18(5):956-62. doi: 10.1200/JCO.2000.18.5.956. PMID 10694544
- [Background] Vardiman JW, Thiele J, Arber DA, Brunning RD, Borowitz MJ, Porwit A, Harris NL, Le Beau MM, Hellstrom-Lindberg E, Tefferi A, Bloomfield CD. The 2008 revision of the World Health Organization (WHO) classification of myeloid neoplasms and acute leukemia: rationale and important changes. Blood. 2009 Jul 30;114(5):937-51. doi: 10.1182/blood-2009-03-209262. Epub 2009 Apr 8. PMID 19357394
- [Background] Garcia-Manero G, Estey EH, Jabbour E, et al. Phase II Study of 5-Azacitidine and Vorinostat in Patients (pts) with Newly Diagnosed Myelodysplastic Syndrome (MDS) or Acute Myelogenous Leukaemia (AML) not eligible for Clinical Trials because of poor performance or presence of other comorbidities. Blood (ASH annual meeting abstracts) 116: Abstract 604, 21010.
- [Background] Guieze R, Jouinot A, Itzykson R, et al. Azacytidine (AZA) in Relapsed MDS and AML after allogeneic stem cell transplantation (allo-HSCT): Results of the French ATU Program. Blood (ASH Annual Meeting Abstracts), Abstract 1293, 2010.
- [Background] Craddock C, Goardon N, Griffiths M, et al. 5' Azacitidine in combination with Valproic Acid induces complete remissions in patients with advanced Acute Myeloid Leukaemia but does not eradicate clonal leukaemic stem/progenitor cells. Blood (ASH Annual Meeting Abstracts), 112: Abstract 945, 2008.
- [Background] Craddock CF, Goardon N, Quek L. et al. 5'azacitidine in combination with valproic acid induces complete remissions in patients with advanced acute myeloid leukaemia but does not eradicate clonal leukaemic progenitors. Blood (ASH annual meeting abstracts), Abstract 638, 2011.
- [Background] Silverman LR, Verma A, Odchimar-Reissig R et al. A Phase I Trial of the Epigenetic Modulators Vorinostat, in combination with Azacitidine (azaC) in Patients with the Myelodysplastic Syndrome (MDS) and Acute Myeloid Leukaemia (AML): A Study of the New York Cancer Consortium. Blood (ASH Annual Meeting Abstracts), 112: Abstract 3656, 2008.